CLINICAL TRIAL: NCT01757067
Title: EVAC-HF is a Prospective, Multi-center, Randomized Study to Compare the Effects on LV Systolic Function Following Radiofrequency Catheter Ablation of Frequent Premature Ventricular Contraction With Optimized Medical Therapy Alone.
Brief Title: Early Elimination of Premature Ventricular Contractions in Heart Failure
Acronym: EVAC-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit sufficient participants
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Timm-Michael Dickfeld, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00053625
Record Dates: First submitted 2012-12-03; First posted 2012-12-28 (Estimated); Results first posted 2021-02-15 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-02

CONDITIONS: Premature Ventricular Contractions; Congestive Heart Failure
Keywords: ablations; CHF; PVC
MeSH Terms: conditions — Ventricular Premature Complexes; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ablation procedure vs medical therapy (Active Comparator): PVC ablation vs medical therapy
  Interventions: Device: PVC ablation
- Compare 2 arms for safety, symptoms (No Intervention): Compare control of PVC's between 2 groups.

INTERVENTIONS:
Device: PVC ablation — This will compare symptoms, safety between ablation procedure vs medical therapy. Biosense Catheter used is not indicated specifically for PVC ablations and will be evaluated
  Other Names: Surround Flow ablation catheters- Biosense Webster
  Arms: ablation procedure vs medical therapy

SUMMARY:
Premature ventricular contractions (PVC) are a very common irregular heart beat (arrhythmias) even in patients without heart disease. Frequent PVCs are thought to occur in about 1-4% of the general population. Many patients with PVCs complain about skipping of their heart (palpitations), shortness of breath and feeling tired. In some patients PVCs may also result in weakening of the heart muscle (heart failure), which might be reversible with suppression of the PVCs.

DETAILED DESCRIPTION:
A common way to get rid of PVCs is an ablation procedure during which a small area of heart muscle that creates the PVCs is cauterized, so that it can no longer cause PVCs. This has been performed for many years and is an overall safe and effective procedure to eliminate PVCs. In the ablation, a catheter with an electrode at its tip is guided with moving X-rays (fluoroscopy) displayed on a video screen to the exact site inside the heart where cells give off the electrical signals that stimulate the abnormal heart rhythm. Radiofrequency energy (similar to microwave heat) is transmitted from the catheter tip to the area. This destroys carefully selected heart muscle cells in a very small area (about 1/5 of an inch) and can stop the area from creating the extra impulses that cause the extra heartbeats. Additionally, some medications have the ability to suppress PVCs (antiarrhythmic medications). PVC ablation and antiarrhythmic medications have both been used to treat patients with PVC's and a reduced heart function. The heart function is referred to as ejection fraction (measured by cardiac ultrasound (echocardiogram). In this study it will be required the ejection fraction will be less than less than or equal to 45% (with 55% or more being normal).

If enrolled in the study there is a 50/50 chance (like a coin toss and referred to as randomization) that the patient will either continue on the best currently available medical treatment for a weak heart muscle (as determined by the doctor) or will undergo a PVC catheter ablation (with a possible second ablation or antiarrhythmic medication, if the first ablation was not a success).

All patients in the study will continue to take the best possible medications for the heart muscle weakness. If the patient is randomized to not undergo the ablation they will be monitored and at the end of 6 months of participation may choose to have the PVC ablation. If a deterioration may occur patients in the control group can have an ablation earlier.

ELIGIBILITY:
Inclusion Criteria:

* Patients with reduced ejection fraction (EF ≤45%) demonstrated by transthoracic echocardiogram and deemed to be non-ischemic by nuclear stress test or cardiac catheterization.
* Patients with >20% PVCs on 24 hour holter-recording
* Patient is 18 years of age or older
* Optimized medical therapy on stable therapy for minimum 3 months with no changes in beta-blocker, ACE-I/ARB, digoxin doses (varying diuretic doses permitted).

Exclusion Criteria:

* Patients who are under the age of 18 years of age
* Patients with >2 dominant PVC morphologies
* Patients with cardiac surgery in previous 3 months or scheduled for following 6 months
* Patients who were implanted with a biventricular device during the last three months or single/dual chamber device (with ventricular pacing >10%) during the last three months
* Significant symptoms associated with PVCs that would make favor immediate ablation
* Intracardiac mural thrombus or myxoma
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-01; Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timm Dickfeld, MD, Principal Investigator — University of Maryland, College Park
Locations (8):
- United States (7):
  - UCLA, Los Angeles, California
  - University of Maryland Medical Center, Baltimore, Maryland
  - University maryland medical Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
- University of Quebec, Sainte-Foy, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PVC Ablation Plus Optimal Medical Therapy: Patients will receive optimal medical therapy including beta blocker or afterload reduction with e.g. ACE-inhibitors as directed by treating local cardiologist/electrophysiologist.
  In addition patient will undergo radiofrequency ablation of PVC guided by current gold standard of ablation including pace mapping and activation mapping to reduce the PVC burden.
- Optimal Medical Therapy: Patients will receive optimal medical therapy including beta blocker or afterload reduction with e.g. ACE-inhibitors as directed by treating local cardiologist/electrophysiologist.
Period: Overall Study
Arm/Group | PVC Ablation Plus Optimal Medical Therapy | Optimal Medical Therapy
Started (The study was closed due to low enrollment.) | 2 | 1 (The study was closed due to low enrollment.)
Completed (The study was closed due to low enrollment.) | 2 (The study was closed due to low enrollment.) | 1 (The study was closed due to low enrollment.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The site enrolled 3 participants in the study
Groups:
- Ablation Procedure: Patient received PVC ablation in addition to optimal medical therapy
- Medical Therapy: Optimal medical therapy
- Total: Total of all reporting groups
Arm/Group | Ablation Procedure | Medical Therapy | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67 (3) | 68 (0) | 67 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 0 | 1
  Canada | 1 | 0 | 1
  China | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change of Left Ventricular Ejection Fraction Measured With Simpson's Rule Expressed in Percent From Pre to Post Intervention
Description: Left ventricular ejection fraction with Simpson's Rule. This is a measurement obtained on an echocardiogram. It reflects the percentage of blood that is ejected from the heart with each beat. The mean change in ejection fraction will be compared for the 2 groups
Time Frame: Change between 0 and 6 months
Population: Due to very low enrollment and closure of study no meaningful statistical analysis could be performed
Measure: Mean (Standard Deviation); unit: Percentage of EF
Groups:
- Ablation Procedure: PVC ablation will be performed in these patients in addition to optimal medical therapy.
- Optimal Medical Therapy: group received only optimal medical therapy
Arm/Group | Ablation Procedure | Optimal Medical Therapy
Number analyzed (Participants) | 2 | 1
Percentage of EF | 35 (5) | 30
Statistical Analysis 1: Comparison: Ablation Procedure vs Optimal Medical Therapy; Test type: Other — The previously stated primary and secondary endpoints cannot be calculated as the study was halted prematurely due to lack of enrollment. Only the reported EF data was collected. This makes further statistical analyses impossible; The previously stated primary and secondary endpoints cannot be calculated as the study was halted prematurely due to lack of enrollment. Only the reported EF data was collected. This makes further statistical analyses impossible

ADVERSE EVENTS:
Time Frame: 0 to 6 months
Groups:
- Ablation Procedure and Optimal Medical Therapy: In the group that received PVC ablation and optimal medical therapy no AE occured.
- Optimal Medical Therapy: In the group that received optimal medical therapy no AE occured
Arm/Group | Ablation Procedure and Optimal Medical Therapy | Optimal Medical Therapy
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2011-09-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT01757067/Prot_000.pdf
  • Statistical Analysis Plan (2011-09-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT01757067/SAP_001.pdf
  • Informed Consent Form (2015-10-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT01757067/ICF_002.pdf